CLINICAL TRIAL: NCT01767337
Title: Exploratory Evaluation of Healthy Subjects Receiving Varied Dose Volumes of Saline Delivered by a Non-Significant Risk Investigational Device Utilizing a Micro-Needle Array
Brief Title: Intracutaneous Delivery of Varied Dose Volumes of Saline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FluGen Inc (Industry)
Collaborators: Accelovance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FGN-NSR-2012-002
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Influenza
Keywords: microneedle-based delivery; hollow microneedle; intracutaneous; drug delivery
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- injection of 0.1 mL saline (Experimental): deliver from FluGen 101.2 device
  Interventions: Device: FLUGEN 101.2 device
- injection of 0.25 mL saline (Experimental): deliver from FluGen 101.2 device
  Interventions: Device: FLUGEN 101.2 device
- Injection of 0.5 mL saline (Experimental): deliver from FluGen 101.2 device
  Interventions: Device: FLUGEN 101.2 device

INTERVENTIONS:
Device: FLUGEN 101.2 device
  Other Names: FLUGEN 101.2

SUMMARY:
This study will evaluate intracutaneous delivery of 0.1, 0.25 and 0.5 milliliter volumes of saline from the FLUGEN 101.2 investigational microneedle-based device.

DETAILED DESCRIPTION:
An intracutaneous delivery device will be evaluated for ability to inject various volumes of saline into subjects skin.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and/or understand and sign the Informed Consent form

Exclusion Criteria:

* Medical history of acute or chronic skin disease
* Active skin allergy or acute skin infection, presence of tattoo(s), scars, sunburn or skin abnormalities at any prospective injection site
* Hirsute at any prospective injection site
* Diabetes
* High levels of anxiety or depression or history of psychosis
* Abuse of alcohol or use of other drugs of abuse including tobacco
* Pregnant or breastfeeding women
* Any medical condition that may interfere with study protocol adherence including completion of study activities
* Foreseeable inability to complete the study as scheduled.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the safety and tolerability/reactogenicity of various saline volumes delivered from the FLUGEN 101.2 microneedle-based device as evidenced by change of dose site appearance over time. | 30 minutes, 24 hours, ~ 1 week
  Observe injection sites for change of appearance post-dose including initial wheal formation and subsequent resolution.

SECONDARY OUTCOMES:
A secondary objective of this study is to evaluate the mechanical elimination of fluid from the device. | 3 minutes
  Evaluate ability of device to dispense targeted dose volume.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Herber, Study Director — FluGen Inc; Murray A Kimmel, DO, Principal Investigator — Accelovance
Locations (1):
- Accelovance Inc, Melbourne, Florida, United States

IPD SHARING:
Plan to Share IPD: No